CLINICAL TRIAL: NCT06623799
Title: Impact of Help-Seeking Behaviors on Allergic Rhinitis, Asthma Control, and Mental Health: A Retrospective and Longitudinal Analysis of Allergy Medication Use
Brief Title: Impact of Help-Seeking Behaviors on Allergic Rhinitis and Mental Health: A Longitudinal Study
Status: Recruiting | Type: Observational
Sponsor: QHSLab, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: QHSLab 001-2024
Record Dates: First submitted 2024-09-13; First posted 2024-10-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Conditions; Allergic
Keywords: Allergic Rhinitis; Asthma Control; Mental Health; Help-Seeking Behaviors; Integrated Care
MeSH Terms: conditions — Rhinitis, Allergic; Psychological Well-Being; Help-Seeking Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study explores how help-seeking behaviors for both emotional well-being and allergies impact the management of allergic rhinitis, asthma, and mental health symptoms, including anxiety and depression. The research involves a retrospective and longitudinal analysis of patients who sought treatment for allergic rhinitis and mental health concerns. The goal is to highlight the importance of integrating mental health care into allergy treatment plans to improve overall patient outcomes.

DETAILED DESCRIPTION:
This study aims to investigate the impact of help-seeking behaviors (HSB) on allergic rhinitis (AR), asthma control, and mental health outcomes, such as anxiety and depression, using both retrospective and longitudinal data. The study examines patients who have been diagnosed with AR and mental health conditions to assess how seeking professional help for allergies, emotional well-being, or both influences symptom control and quality of life.

The research analyzes data from a diverse patient population to evaluate the effects of AR medications (intranasal steroids, antihistamines, decongestants, and leukotriene blockers) on both AR and mental health symptoms. Additionally, it explores the role of help-seeking behaviors in improving symptom management, specifically through the use of validated tools like the SNOT-22 for AR and the PHQ-GAD16 for mental health.

The study emphasizes the importance of integrating mental health screening and support into the treatment of allergic rhinitis and asthma. By analyzing real-world data, the research seeks to provide insights into how coordinated care approaches can enhance patient outcomes and inform future clinical practices.

ELIGIBILITY:
Inclusion Criteria:

Adults (aged 18 years or older) Patients actively receiving care in a primary care setting. Patients who have provided informed consent for their health data to be included in the research repository.

Exclusion Criteria:

Patients who have not provided informed consent for their health data to be included in the research repository.

Patients diagnosed with chronic conditions outside the scope of allergic rhinitis, asthma, or mental health conditions (anxiety, depression).

Patients with severe mental health disorders or comorbidities that are unrelated to the conditions of interest (e.g., schizophrenia, bipolar disorder, etc.).

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This repository collects data from primary care patients diagnosed with allergic rhinitis, asthma, anxiety, or depression. The repository aims to track health outcomes, medication usage, and help-seeking behaviors to support future research on the interaction between chronic physical and mental health conditions. The population includes adult patients who consent to the inclusion of their data and who seek care in a primary care setting for the specified conditions.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Change in Allergic Rhinitis Symptom Severity (SNOT-22 Score) | baseline and yearly follow-up for up to 5 years
  This outcome measures the long-term change in allergic rhinitis symptom severity over several years using the Sinonasal Outcome Test (SNOT-22). The SNOT-22 is a validated tool that assesses the impact of sinonasal conditions on quality of life. The study will track the effects of help-seeking behaviors for both allergies and mental health (anxiety and depression) on allergic rhinitis symptom control, examining changes in SNOT-22 scores over multiple follow-up periods. Scores range from 0 to 110, with higher scores indicating worse symptoms and lower quality of life.

SECONDARY OUTCOMES:
Change in Depression Symptoms (PHQ-9 Score) | Baseline and yearly follow-up for up to 5 years
  This outcome measures the change in depressive symptoms using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a validated tool to assess the severity of depression. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. The study will assess how help-seeking behaviors for both allergies and mental health impact the severity of depressive symptoms over time.
Change in Anxiety Symptoms (GAD-7 Score) | Baseline and yearly follow-up for up to 5 years
  This outcome measures the change in anxiety symptoms using the Generalized Anxiety Disorder Scale (GAD-7). The GAD-7 is a validated tool to assess the severity of anxiety. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. The study will assess how help-seeking behaviors for both allergies and mental health impact the severity of anxiety symptoms over time.

OTHER OUTCOMES:
Effect of Help-Seeking Behaviors on Symptom Control and Quality of Life | Baseline and yearly follow-up for up to 5 years
  This outcome evaluates the effect of help-seeking behaviors (seeking help for emotional well-being, allergies, or both) on overall symptom control and quality of life. The study will explore the relationship between help-seeking behaviors and improvements in allergic rhinitis symptoms (SNOT-22) and mental health outcomes (PHQ-9, GAD-7). Scores from each scale will be analyzed separately to assess the impact of help-seeking behaviors on these specific health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- QHSLab, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the need to protect patient confidentiality. Data collected in this study is used for internal analysis, and only aggregated, anonymized data will be made available for research purposes. This ensures compliance with privacy regulations such as HIPAA and protects patient identities.